CLINICAL TRIAL: NCT04527523
Title: Incidence of Post-operative Cystoid Macular Edema: A Prospective Study Comparing DMEK, DSEK, and DSO
Brief Title: Descemet Membrane Endothelial Keratoplasty vs. Descemet's Stripping With Endothelial Keratoplasty vs. Descemet Stripping Only
Status: Terminated | Type: Observational
Why Stopped: PI does not have the time and support needed to continue the study at this time.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00067948
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cystoid Macular Edema; Fuchs Dystrophy
Keywords: endothelial transplants; endothelial dysfunction
MeSH Terms: conditions — Macular Edema; Fuchs' Endothelial Dystrophy | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endothelial Dysfunction Cohort: All patients enrolled in the study will receive a baseline Optical Coherence Tomography scan (OCT) within 4 weeks prior to surgery. Two additional OCT scan will be performed 6 weeks and 3 months after surgery.
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — OCT is an imaging method that uses light waves to create images of the retina.
  Other Names: OCT

SUMMARY:
This study aims to evaluate and compare incidence of post-operative cystoid macular edema (CME) after Descemet Membrane Endothelial Keratoplasty (DMEK), Descemet's Stripping Automated endothelial Keratoplasty (DSEK) and Descemet Stripping Only (DSO).

DETAILED DESCRIPTION:
Patients that are undergoing any of these procedures will be asked if they are willing to have a baseline pre-operative Optical Coherence Tomography (OCT) scan completed within 4 weeks of surgery. Additional OCT scans will be collected during routine follow up care. It is hypothesized that the rates of CME will be lower with DSO compared to DMEK and DSEK.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that is undergoing DSO or endothelial corneal transplantation vis DMEK or DSEK

Exclusion Criteria:

* Patients that do not have an optical coherence tomography measurement pre- operatively
* Patients that don't have an optical coherence tomography measurement post- operatively
* Patients with a previous history of uncontrolled macular edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endothelial dysfunction that require treatment, and are being evaluated for Descemet Stripping Only (DSO), Descemet Membrane Endothelial Keratoplasty (DMEK) or Descemet's Stripping Automated Endothelial Keratoplasty (DSEK)
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-Op CME | 6 weeks post-operative
  The frequency (number of Subjects) of post-operative Cystoid Macular Edema will be evaluated for patients receiving DMEK, DSEK or DSO.
Incidence of Post-Op CME | 3 months post-operative
  The frequency (number of Subjects) of post-operative Cystoid Macular Edema will be evaluated for patients receiving DMEK, DSEK or DSO.
Severity of Post-Op CME | 6 weeks post-operative
  The severity of post-operative Cystoid Macular Edema will be evaluated for patients receiving DMEK, DSEK or DSO that experience Cystoid Macular Edema after surgery - measured by net change of Central Foveal Thickness on Optical Coherence Tomography (OCT- is an imaging technique that uses low-coherence light to capture micrometer-resolution, two- and three-dimensional images from within optical scattering media, e.g., biological tissue)
Severity of Post-Op CME | 3 months post-operative
  The severity of post-operative Cystoid Macular Edema will be evaluated for patients receiving DMEK, DSEK or DSO that experience Cystoid Macular Edema after surgery - measured by net change of Central Foveal Thickness on Optical Coherence Tomography (OCT- is an imaging technique that uses low-coherence light to capture micrometer-resolution, two- and three-dimensional images from within optical scattering media, e.g., biological tissue)

SECONDARY OUTCOMES:
Graft Detachment | 6 weeks and 3 months post-operative
  Frequency (number of Subjects) of post-operative graft detachment will be evaluated in patients that receive a corneal endothelial transplant.
Re-bubbling Procedure | 6 weeks and 3 months post-operative
  The incidence (number of Subjects) of re-bubbling procedures performed post-operatively will be evaluated.
Infection | 6 weeks and 3 month post-operative
  The incidence (number of Subjects) of post-operative infection will be evaluated.
Final Visual Acuity | 3 months post-operative
  The Snellen Visual Acuity test - This means that the test subject sees the same line of letters at 20 feet that person with normal vision sees at 20 feet. 20/40 vision means that the test subject sees at 20 feet what a person with normal vision sees at 40 feet.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Giegengack, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. Final, overall results will be reported for each outcome.

REFERENCES:
- [Background] Inoda S, Hayashi T, Takahashi H, Oyakawa I, Yokogawa H, Kobayashi A, Kato N, Kawashima H. Risk Factors for Cystoid Macular Edema After Descemet Membrane Endothelial Keratoplasty. Cornea. 2019 Jul;38(7):820-824. doi: 10.1097/ICO.0000000000001950. PMID 30973407
- [Background] Kocaba V, Mouchel R, Fleury J, Marty AS, Janin-Manificat H, Maucort-Boulch D, Burillon C. Incidence of Cystoid Macular Edema After Descemet Membrane Endothelial Keratoplasty. Cornea. 2018 Mar;37(3):277-282. doi: 10.1097/ICO.0000000000001501. PMID 29298168
- [Background] Arbelaez JG, Price MO, Price FW Jr. Long-term follow-up and complications of stripping descemet membrane without placement of graft in eyes with Fuchs endothelial dystrophy. Cornea. 2014 Dec;33(12):1295-9. doi: 10.1097/ICO.0000000000000270. PMID 25299425
- [Background] Koenig SB. Planned Descemetorhexis Without Endothelial Keratoplasty in Eyes With Fuchs Corneal Endothelial Dystrophy. Cornea. 2015 Sep;34(9):1149-51. doi: 10.1097/ICO.0000000000000531. PMID 26186374